CLINICAL TRIAL: NCT03347799
Title: WINROP Algorithm Validation for Retinopathy Screening in Premature Infants: a Retrospective Cohort Analysis Over 4 Years
Brief Title: WINROP Algorithm Validation for Retinopathy Screening in a Cohort of Premature Infants
Acronym: WINROP
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Michel HASCOET, Professor, Central Hospital, Nancy, France
Other Study IDs: PSS2016/WINROP-HASCOET/VS
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Retinopathy of Prematurity
Keywords: very premature infants; screening; retinopathy
MeSH Terms: conditions — Retinopathy of Prematurity; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
When a child was born too early, it is more likely to develop an alteration of its visual function than in the case of term birth. Significant visual disturbances are found in 3% of children born prematurely, but visual impairment can be very severe, up to the loss of vision in case of retinopathy of prematurity (ROP) in the most immature infants. The introduction of screening surveillance systems, such as WINROP software, might reduce the need for stressful eye examination in low risk neonates. This retrospective study aimed at validating the WINROP algorithm in a cohort of premature infants, born below 32 weeks of gestation, who had systematic eye examination for ROP screening over 4 year period.

ELIGIBILITY:
Inclusion Criteria:

* All infants born below 32 weeks gestation within the study period
* At least one eye examination recorded by Retcam

Exclusion Criteria:

* Any ophthalmic abnormality
* Any genetic abnormality

Ages: 24 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants, born from July 2012 to July 2016, from 24 to 32 weeks gestation had hospitalized in our level III NICU having had eye examination up to 40 weeks post menstrual age.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
algorithm validation | from birth up to 40 weeks post menstrual age
  risk of retinopathy occurence

SECONDARY OUTCOMES:
risk factor for retinopathy | from birth up to 40 weeks post menstrual age
  standardized perinatal data collection

IPD SHARING:
Plan to Share IPD: No